CLINICAL TRIAL: NCT03389516
Title: Healing Nipple Wounds: Comparison Between 2 Treatment Modalities: Lanolin Ointmentnad Nursicare Therapeutic Breast Pads Among Postpartum Mothers Dealing With Sore Nipples
Brief Title: Healing Nipple Wounds: Comparison Between 2 Treatment Modalities
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laniado Hospital (Other)
Collaborators: Dr. Jinna Weissman (Unknown)
Responsible Party: Principal Investigator, Dr. Meir Weisbrod, Director of Neonatal Department, Laniado Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0142-16-LND
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Nipple Wounds
MeSH Terms: interventions — Polymem; Lanolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polymem breast pads (Active Comparator)
  Interventions: Other: Polymem
- Lanolin (Active Comparator)
  Interventions: Other: Lanolin

INTERVENTIONS:
Other: Polymem — wound care dressings
  Other Names: Nursicare
  Arms: Polymem breast pads
Other: Lanolin — wound care oinment
  Other Names: Lansinoh
  Arms: Lanolin

SUMMARY:
It is widely accepted that breast milk is the optimal source of infant nutrition. Despite the World Health Organization (WHO) recommendation of exclusive breastfeeding for the first 6 months of infant life, many women discontinue breastfeeding as a result of perceived difficulties. In Israel, 88.4% of mothers declare about their intentions to breastfeed. Only 70.9% are still breastfeeding 2 months postpartum. Nipple pain is a highly prevalent, significant reason for breastfeeding cessation.

In the past, we encouraged wound healing nipples by drying (air drying; sun; other heat source). It turned out that this drying only delays the healing due to lack of moisture, causing cracks in the outer layer of the nipple. Today, nipple wound care needs treatment approaches consistent with wounds treatment in other body parts (moist wound healing), and which also addresses reduction of pain. Studies have shown that the preservation of moisture accelerates healing and allows epithelization.

In the past couple of years, the Nursicare therapeutic breastfeeding pads have become a commonly used option for sore nipples. Nursicare pads enhance moist wound healing and soothe traumatized tissues, localize the inflammation, reducing wound pain and providing comfort at the wound site. This solution seems to be more efficient, and pads can be removed with virtually no pain and no remnants on the nipple that might cause concerns for allergic reaction for the infant.

In this clinical trial we attempt to compare between the 2 treatments: Lanolin ointment and Nursicare therapeutic breast pads among postpartum mothers dealing with sore nipples and to examine the effectiveness of each treatment for short term (period till primary pain relief) and long term (total period for wound closure).

Study hypothesis is that Nursicare provides better pain relief and faster healing that Lanolin.

Method The trial will include postpartum mothers in Laniado Hospital in Natanya and mother from "Halav M" breastfeeding clinic in Olesh, Israel who had complained of nipple pain with any sign of nipple trauma to one or both nipples.

The participants will be randomly selected to each group:

1. Treatment with the Nursicare therapeutic breastfeeding pads.
2. Treatment with application of Lanolin. A total number of participants: At least 50 mothers randomly chosen to each group will be recruited for this trial (p). Randomization will be based on natural arrival sequence - where every other mother will be placed on 'Nursicare group' and the alternate every other mother will be placed in 'control/Lanoline group). The only exception for this is when a certain treatment is already started - in those cases the patient will continue that treatment and compensation will be done to the sequence of allocation process.

DETAILED DESCRIPTION:
It is widely accepted that breast milk is the optimal source of infant nutrition. Despite the World Health Organization (WHO) recommendation of exclusive breastfeeding for the first 6 months of infant life, many women discontinue breastfeeding as a result of perceived difficulties. In Israel, 88.4% of mothers declare about their intentions to breastfeed. Only 70.9% are still breastfeeding 2 months postpartum. Nipple pain is a highly prevalent, significant reason for breastfeeding cessation.

Sore nipples or breast is indeed one of the common problems during breastfeeding but it is difficult to define its incidence accurately. Literature reports on the frequency of nipple pain range from: A majority of mothers reporting painless breastfeeding at 6 days postpartum [1] to reports of pain in 96% of all breastfed women in the first 6 weeks after birth [2]. The reasons for the wide variation in pain reporting are that the perception of pain is subjective, and also because there is a great deal of methodological difference in studies of nipples and breast pain.

Sore nipples or breast are considered one of the main reasons for discontinuation of breastfeeding [3, 4, 5, 6, 7]. With about 30% of mothers suffering from pain and nipple lesions may switch to other feeding methods within 6 weeks [7]. Even when there is no premature weaning, the mother's breastfeeding experience is impaired, and the mother-infant relationship may be damaged [8, 9]. In addition, it was reported that pain in breastfeeding harms the quality of sleep, the activities and mood of the mother [10].

Although breast pain is a common condition, it can be prevented and treated. It is important to distinguish between physiological sensitivity and pain. In case of tenderness during breastfeeding, the nipple will appear normal and round at the end of the feeding, and it should pass within 2-3 days without the development of clinical signs of injury. The source of the sensitivity is probably hormonal or arises mostly from the negative pressure exerted on the milk ducts before they are filled with milk [11]. When it comes to pain that lasts longer than two days and is accompanied by a worsening, or there are signs of injury to the breast from the beginning, the common cause is an incorrect latch of the nipple in the baby's mouth. In this case, it is essential to correct the technique as the main part of the treatment required.

There are several common treatments among mothers for sore nipples. The 2 most frequently used are:

1. Lanolin
2. Breast milk In the past, we encouraged wound healing nipples by drying (air drying; sun; other heat source). It turned out that this drying only delays the healing due to lack of moisture, causing cracks in the outer layer of the nipple. Today, nipple wound care needs treatment approaches consistent with wounds treatment in other body parts (moist wound healing), and which also addresses reduction of pain. Studies have shown that the preservation of moisture accelerates healing and allows epithelization.

In the past couple of years, the Nursicare therapeutic breastfeeding pads have become a commonly used option for sore nipples. As in other PolyMem® products, that enhance moist wound healing and soothes traumatized tissues, localize the inflammation, reducing wound pain and providing comfort at the wound site, I can see the same effect in my clinical experience with Nursicare therapeutic breastfeeding pads while treating nipple wounds. This solution seems to be more efficient, and pads can be removed with virtually no pain and no remnants on the nipple that might cause concerns for allergic reaction for the infant.

In this clinical trial we attempt to compare between the 2 treatments: Lanolin ointment and Nursicare therapeutic breast pads among postpartum mothers dealing with sore nipples, and to examine the effectiveness of each treatment for short term (period till primary pain relief) and long term (total period for wound closure).

Study hypothesis is that Nursicare provides better pain relief and faster healing that Lanolin.

Method The trial will include postpartum mothers in Laniado Hospital in Natanya and mother from "Halav M" breastfeeding clinic in Olesh, Israel who had complained of nipple pain with any sign of nipple trauma to one or both nipples.

The participants will be randomly selected to each group:

1. Treatment with the Nursicare therapeutic breastfeeding pads.
2. Treatment with application of Lanolin. A total number of participants: At least 50 mothers randomly chosen to each group will be recruited for this trial (p). Randomization will be based on natural arrival sequence - where every other mother will be placed on 'Nursicare group' and the alternate every other mother will be placed in 'control/Lanoline group). The only exception for this is when a certain treatment is already started - in those cases the patient will continue that treatment and compensation will be done to the sequence of allocation process.

The first 10-14 mothers will constitute a pilot. After data collection among at least five participants in each group we will validate the questionnaire and the collected data to secure that our processes and protocols are as intended. This should be seen as a pilot study integrated in the overall study design. This pilot/validation process will hopefully confirm that our processes are in line with research objective - and we will continue study. Worst case, if we discover significant flaws we will have to restart the data collection process after tuning our protocols.

The data collection will take place in different time points and ways:

Time points:

1. Zero point:

   1. Pain level collected at start of session
   2. Complete questionnaire filled in (Approx. 30 min) + picture if possible
2. At the end of the questioner session - Approx. 30 minutes: Pain level collected
3. During the first 4-6 hours after applying the treatment - pain level collected (by phone call or interactive questionnaire)
4. 24 hours after applying the treatment - questionnaire by phone call or interactive questionnaire
5. 3 days after applying the treatment - Second meeting will take place in the breastfeeding clinic "Halav M" or in the maternity ward in Laniado Hospital.
6. 6 days after applying the treatment - a follow-up third meeting or phone conversation. The option will be examined during the second meeting depends on the conditions of the sore. Third meeting will take place in the breastfeeding clinic "Halav M" or in the maternity ward in Laniado Hospital. In any case a questionnaire will be filled after 6 days.
7. A follow up by phone calls will be carried out till full wound closure on days: 14 and 30.

In each phone call / interactive questionnaire, the mothers will report about their pain, comfort, breastfeeding issues, etc.

In each meeting (including the first one), the sores and pain will be examined by the following methods:

1. Sore and nipple condition and secretions will be examined by the tester
2. VAS scale ruler by the mother
3. VAS scale ruler by the tester
4. Stage of nipple trauma (Mohrbacher scale, 2004)
5. Size of the wound surface (mm2) The key endpoints that will be exanimated are: (measurement in brackets)

   * Pain reduction (VAS scale)
   * Improvement in wound closure (percentage of wounds closed at each measure point - 3 days & 6 days)
   * Status of wound closure: (staging at each measure point)
   * Transition to full breastfeeding (Measurement to be filled in the questioner)
   * Product satisfaction (Very unhappy - unhappy - neutral - happy - very happy)
   * Ease of use (Very troublesome - troublesome - neutral - easy - very easy)
   * Recommendation to others (Would you recommend this product to your best friend? No - Not sure - Yes(
   * The response for future use if necessary (Would you be happy to use this product again? No - Not sure - Yes)

The data will be analyzed and processed using SPSS version 22 software. Between-group differences (Lanolin vs Nursicare) for dichotomous outcome data will be analyzed by χ2 test and for continuous data by t test.

Survival analysis model will be used to estimate the time to wound closure. If necessary, tests will be carried out nonparametric analysis. For all test results P≤ 0.005 will be considered statistically significant. The statistical error expected to be 10%.

The clinical and statistical results will be presented.

ELIGIBILITY:
Inclusion Criteria:

Postpartum breastfeeding mothers for healthy babies, who will meet the following inclusion criteria:

Maternal complaint of nipple pain with any sign of nipple trauma to one or both nipples, such as blistering, crusting, redness, bleeding, swelling, cracking, discoloration or peeling caused by breastfeeding or pumping.

-

Exclusion Criteria:

Mothers having the following will be excluded from the study:

* Mothers with diabetes (it is known that diabetes impacts on wound healing and to avoid any credibility questions linked to this it is considered prudent to leave mothers with diagnosed diabetes out of the study)
* Mothers with skin allergies or taking medications for skin allergies
* Psychiatric patients who cannot give consent
* Mothers with grade IV nipple sores
* Mothers with skin diseases:

  * thrush
  * Stephen Johnson Disease
  * Psoriasis
  * Pampigos

Mothers who will not undergo the full clinical follow-up program and will not arrive for at least one follow-up meeting will be excluded from the study.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | • zero point • 30 minutes after applying the treatment • 4-6 hours after applying the treatment • 24 hours after applying the treatment • 3 days after applying the treatment • 6 days after applying the treatment
  VAS scale will be used at several time points in order to assess the duration of pain reduction:
  1. VAS scale ruler by the mother - if zero represents no pain and ten represents the worst pain imaginable, what number best describes the pain you have?
  2. VAS scale ruler by the tester - If zero represents no pain and ten represents the worst pain imaginable, what number best describes the pain you think the mother has?
Wound improvement | • zero point • 3 days after applying the treatment • 6 days after applying the treatment (only in case the meeting will take place, according to the decision taken on day 3)
  measurement of the percentage of wounds closed at each measure point. We will calculate the surface of the wound using an application for calculating area or with a disposable tape measure from paper.

SECONDARY OUTCOMES:
Transition to full breastfeeding | • zero point • 30 minutes after applying the treatment • 4-6 hours after applying the treatment • 24 hours after applying the treatment • 3 days after applying the treatment • 6 days after applying the treatment
  This measurement will be filled in the questioner:
  How do you feed your baby today?
  1. Breastfeeding only
  2. Breastfeeding combined with something else
Product satisfaction | At follow up by phone calls on days: 14 and 30.
  This measurement will be filled in the questioner:
  Were you satisfied with the use of Nursicare®/Lanolin as a treatment to your nipple pain?
  1. Very satisfied
  2. Satisfied
  3. Moderately satisfied
  4. Not satisfied
  5. Not satisfied at all
  6. It didn't affect me
Ease of use | At follow up by phone calls on days: 14 and 30.
  This measurement will be filled in the questioner:
  How did you find Nursicare® pads/Lanolin convenient to use?
  1. Very convenient
  2. Convenient
  3. Not convenient
  4. Not convenient at all
Recommendation to others | At follow up by phone calls on days: 14 and 30.
  This measurement will be filled in the questioner:
  Will you recommend your breastfeeding friends toy use Nursicare®/Lanolin in case they have nipple pain?
  1. Definitely yes
  2. Probably yes
  3. I'm not sure
  4. Probably not
  5. Definitely not
The response for future use if necessary | At follow up by phone calls on days: 14 and 30.
  This measurement will be filled in the questioner:
  In case you have another wound in the future, will you use Nursicare®/Lanolin again to treat the pain?
  1. Definitely yes
  2. Probably yes
  3. I'm not sure
  4. Probably not
  5. Definitely not

CONTACTS AND LOCATIONS:
Locations (1):
- Laniado Hospital, The Betty Retter Mother & Baby Medical Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No